CLINICAL TRIAL: NCT03868761
Title: Feasibility and Preliminary Efficacy of a Digital Mental Health Intervention to Reduce Symptoms of Post-Disaster Traumatic Stress, Depression, and Anxiety in Teens Impacted by Wildfires: A Randomized Multiple-Baseline Single-Case Study.
Brief Title: Feasibility and Efficacy of a Digital Mental Health Intervention for Teen Wildfire Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Adrienne Julie Heinz, Research Health Scientist, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-49196
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Disaster; PTSD; Adolescent Behavior; Trauma; Anxiety; Stress
Keywords: Mobile app; Disaster; Digital Medicine; Teens
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Adolescent Behavior; Wounds and Injuries; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, open label non-concurrent multiple-baseline experimental study with participants acting as their own controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): 21 male and female teenage participants will be randomized to one of three varying baseline assessment periods of two, four, or six weeks. Multiple baseline is a type of single-case experimental design (SCED) that is a time- and cost-effective method for evaluating efficacy of a new treatment, Sonoma Rises. The randomization of participants to baseline periods of varying lengths enables assessment of whether symptom changes occur when, and only when, the intervention is applied.
  Interventions: Behavioral: Sonoma Rises

INTERVENTIONS:
Behavioral: Sonoma Rises — All participants will receive the intervention, Sonoma Rises, a mobile app designed by psychologists at the National Center for PTSD for wildfire survivors to facilitate recovery from disaster. Users can access evidence-informed tools to help cope with stress, heal from loss, prioritize self-care, connect with others, manage anger, and track their mood using validated assessments. There are also tools designed just for teens and users are linked to psychoeducation on disaster and health and other mental health resources and services.
  Other Names: Mobile Mental Health App

SUMMARY:
In October, 2017, Northern California experienced devastating and historic wildfires. Sonoma Rises is an app designed for anyone who was impacted by this event and is intended to help survivors of disaster find their new normal. This study will assess the feasibility and efficacy of a self-help post-disaster mental health intervention delivered via a mobile app with a sample of teens who are experiencing post-disaster mental health symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Males & females aged 13-17 years directly impacted by the 2017 wildfires having lost their home or been temporarily displaced
2. Screen positive for PTSD (Child Trauma Screening Questionnaire = 5 or higher)
3. Have regular access to a smart phone and a computer
4. Have a personal email address
5. Speak and read English fluently
6. Have parental consent

Exclusion Criteria:

1. A positive self-reported history of psychosis, bipolar, or schizophrenia
2. Serious self-reported physical health concerns necessitating surgery or with prognosis <6 months
3. A positive screen for a current Substance User Disorder (CRAFFT = 2 or higher)
4. Current self-reported suicidal ideation
5. Self-reported pregnancy
6. Self-reported less than four weeks of stable prescription medication for anxiety, anti-depressant, and sleep promoting medications prior to the screening assessment

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-11-22 (Actual)

PRIMARY OUTCOMES:
Feasibility: intervention retention: number of treatment completers | 4 months
  retention (i.e., number of treatment completers)
Feasibility: intervention safety: number of adverse events | 4 months
  safety (i.e., number of adverse events)
Feasibility: intervention adherence: number of treatment components completed | 4 months
  adherence rates (i.e., number of treatment components completed)
Feasibility: intervention satisfaction/acceptability | 4 months
  satisfaction/acceptability (i.e., participant satisfaction with treatment "how would you rate your overall satisfaction with the program?"- range 0-10 - higher score indicates more satisfaction)
Feasibility: intervention promotion | 4 months
  Net promoter score (i.e., "How likely are you to recommend this to a friend?" score range 0-5; lower score indicates higher likelihood of promotion)
Feasibility: engagement rate | 4 months
  Engagement rate (i.e., Number and average length of logins to the mobile app intervention)
PTSD Symptom Severity | 4 months
  Child PTSD Symptom Scale for Diagnostic and Statistical Manual-5; score ranges from 0-80; higher scores indicate more PTSD symptom severity
PTSD functional impairment | 4 months
  Child PTSD Symptom Scale for Diagnostic and Statistical Manual-5; score ranges from 0-7; higher scores indicate more PTSD related functional impairment

SECONDARY OUTCOMES:
Internalizing symptoms | 4 months
  Behavior and Feelings Survey - Youth; range 0-24; higher scores indicate more internalizing symptoms (anxiety, depression, stress)
Externalizing symptoms | 4 months
  Behavior and Feelings Survey- Youth; range 0-24; higher scores indicate more externalizing symptoms (behavior problems)
Psychosocial functioning | 4 months
  Ohio Youth Scale - Functioning Subscale; Score range 0-80; higher score indicated better functioning

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Heinz, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States